CLINICAL TRIAL: NCT04171856
Title: Exploring Motor Learning in Acute Stroke Through Robotics
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Mont-Godinne (Other)
Responsible Party: Principal Investigator, Pr Yves Vandermeeren, MD, PhD, Principal Investigator, University Hospital of Mont-Godinne
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: B039201938990
Record Dates: First submitted 2019-11-12; First posted 2019-11-21 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Stroke, Acute
Keywords: Acute stroke; Motor skill learning; Upper limb; Rehabilitation; Subacute stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Motor Skill Learning (CIRCUIT) (Experimental): Intervention: training on the REAplan robot with a serious game based on motor skill learning (MSkL) serious game, the CIRCUIT.
  Interventions: Device: REAplan(R)
- Motor control recovery (EASY) (Active Comparator): Training on the REAplan robot with a serious game that requires similar type and amount of movements but does not rely on motor skill learning (EASY), a brick buster game.
  Interventions: Device: REAplan(R)
- Conventional (Active Comparator): Training sessions with classical exercices focused on the upper limb administered by occupation therapist.
  Interventions: Device: REAplan(R)

INTERVENTIONS:
Device: REAplan(R) — motor skill learning with the REAplan(R) rehabilitation robot, to be perfomed with the affected arm

SUMMARY:
The acute phase of stroke is characterized by an enhancement of neural plasticity which supports rapid motor recovery. It is unclear whether acute stroke patients can acquire new motor skills with their affected upper limb. The aims of this research program are:

1. To test the capacity of acute stroke patients (< 21 days) to learn and retain a complex unimanual motor skill.
2. To explore whether acute stroke to different brain regions (quantified with brain MRI) induces specific deficits in motor skill learning.
3. To compare acute stroke patients with healthy individuals and with chronic stroke patients.

DETAILED DESCRIPTION:
Over 3 consecutive days, the subjects will be evaluated and will train on the rehabilitation robot REAplan® (http://www.axinesis.com/). They will practice 2 serious games on the robot.

In order to differentiate the effect of motor control recovery from that of MskL, the acute stroke patients will be randomised 4/1 to "MskL" (n=120) ,to "motor control recovery" (n=30) or to "conventional" group (n=15) with a minimisation software. The experimental design will be similar except that the "motor control recovery" group will practice the serious game EASY instead of CIRCUIT (see below) and the "conventional" group will practice conventional therapy instead of CIRCUIT. The performances on both EASY & CIRCUIT will be compared between groups (subjects in both groups will perform the EASY & CIRCUIT tasks).The total time of rehabilitation will be the same.

The motor skill learning setup (CIRCUIT + EASY) that we developed and successfully used in healthy individuals and stroke patients has already been implemented in the REAplan environment and will be used as innovative serious games based on a speed/accuracy trade-off (SAT), allowing a detailed analysis of motor skill learning components (speed, accuracy, SAT, movement smoothness, dynamics...). For the serious game CIRCUIT, who based on motor skill learning, the subjects will have to practice a complex circuit and move as a cursor quickly and accurately as possible by controlling the handle of the robot with their affected hand/arm. For the other task EASY (a brick busters serious game), the aim will be to go back and forth between walls presented in different locations. The CONVENTIONAL therapy will consist in classical exercices focused in the upper limb administered by occupational therapist.

The subacute stroke phase is a unique opportunity to investigate the role of brain structures in motor learning/control. Compared to chronic impairments (> 6 months post-stroke), the subacute phase provides a window into how a lesion perturbs sensorimotor functions prior to reorganisation driven by plasticity and neurorehabilitation. To clarify the role of different brain structures in MskL, Voxel-based Lesion Symptom Mapping (VLSM) based on high-resolution brain magnetic resonance imaging (MRI) scans, will be used to analyse the relationship between tissue damage and MskL scores on a voxel-by-voxel basis.

In addition, several "classical" clinical scales and tests will be used to evaluate overall motor-sensory-cognitive functions. The subjects will practice serious games on the robot REAplan (R), requiring movements with the affected arm (unimanual tasks).

And, we used a Dextrain® tool which allows quantification of key components of manual dexterity : forces, selectivity (independance of fingers movement) and coactivation of the fingers.Moreover, we added a Transcranial magnetic stimulation (TMS), as a tool for predicting recovery of motor function after stroke.

In addition to the (sub)acute stroke patients, 4 others groups will be recruited for this study : a group of acute stroke patients who will receive "conventional rehabilitation" and be shortly tested on the robot (N=15), a group of chronic stroke patients (stroke > 6 months) who will not be hospitalized and will not undergo MRI (N=30), a group of healthy individuals who will not undergo MRI (N=50) and a group of patients with a transient global amnesia which is a sudden, temporary episode (<24hours) of memory loss (N=15).

Subjects in these 4 groups will be randomized 1/1 in the two arms ("MSkL" versus "motor control recovery" arms), except the patients with a TGA who will be included in the "MSkL" arm only.

ELIGIBILITY:
ACUTE STROKE PATIENTS:

Inclusion Criteria:

* acute stroke (> 21 days)
* aged 18-90 years
* with a stroke lesion on brain imaging

Exclusion Criteria:

* " classical " contre-indication to MRI (non-MR-compatible pacemaker, pregnancy, non-MR-compatible implanted devices, claustrophoby, etc ...)
* difficulty in understanding or executing commands
* drug/alcohol abuse
* severe aphasia / cognitive deficits interfering with study
* inability to voluntarily move the affected arm (i.e. complete paralysis of the arm)
* multiple strokes / dementia / psychiatric condition

PATIENTS WITH TRANSIENT GLOBAL AMNESIA:

Clinical diagnosis, criteria of Hodge & Warlow (1990):

* Anterograde amnesia observed by a witness
* No alteration of consciousness or loss of identity
* Cognitive dysfunction limited to amnesia
* Lack of focused neurological deficit or argument for a comitiality
* Absence of head trauma
* Symptom resolution within 24 hours
* Possible existence of vegetative symptoms

Inclusion criteria:

* Transient global amnesia
* 8-90 years old
* Be able to perform 3 consecutive sessions on a rehabilitation robot

Exclusion criteria:

* Severe aphasia / cognitive deficits interfering with study
* Psychiatric disorders
* Alcohol / drug addiction
* Exclusion criteria related to MRI

HEALTHY INDIVIDUALS:

Inclusion Criteria:

• 18-90 years

Exclusion Criteria:

* medical history with a previous stroke/neurological deficit
* drug/alcohol abuse
* psychiatric condition/ dementia

CHRONIC STROKE PATIENTS:

Inclusion Criteria:

* chronic stroke (>6 months)
* aged 18-90 years
* with a stroke lesion on brain imaging

Exclusion Criteria:

* difficulty in understanding or executing commands
* drug/alcohol abuse
* severe aphasia / cognitive deficits interfering with study
* inability to voluntarily move the affected arm (i.e. complete paralysis of the arm)
* multiple strokes / dementia / psychiatric condition

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 245 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2030-05-01 (Estimated); Study Completion 2040-07-01 (Estimated)

PRIMARY OUTCOMES:
change in SAT (CIRCUIT) | change between Baseline Day1 and Day3 (acute) + between Baseline Day1 and 3/6 and 12 months post-stroke (subacute - chronic)
  Speed/ Accuracy Trade-off
total distance travelled (EASY) | change between Baseline Day1 and Day3 (acute) + between Baseline Day1 and 3/6 and 12 months post-stroke (subacute - chronic)
  total distance travelled between the walls of the brick busters (in cm)

SECONDARY OUTCOMES:
Fugl Meyer Upper Extremity Test | change between Baseline Day1 and Day3 (acute) + between Baseline Day1 and 3/6 and 12 months post-stroke (subacute - chronic)
  Tests impairments of the upper limb after stroke
Arm Motor Ability (AMA) test | change between Baseline Day1 and Day3 (acute) + between Baseline Day1 and 3/6 and 12 months post-stroke (subacute - chronic)
  Measure disabilities of the upper limb after stroke
Fatigue Visual Analog Scale (VAS) | change between Baseline Day1 and Day3 (acute) + between Baseline Day1 and 3/6 and 12 months post-stroke (subacute - chronic)
  Visual Analog Scale to evaluate fatigue between 0 and 10. The maximum value (10) indicate a high level of fatiguability.
Voxel-based Lesion Symptom Mapping (VLSM) | Baseline
  High-resolution 3D-MRI, diffusion MRI (DWI) & perfusion MRI (PWI with Arterial SPin Labelling technique) will be acquired. The stroke areas will be drawn with MRIcron as volumes of interest (VOI) in native space and compared.
Dextrain® | change between Baseline Day1 and Day3 (acute) + between Baseline Day1 and 3/6 and 12 months post-stroke (subacute - chronic)
  Quantitative assessment of the manual dexterity : fingers strength and selectivity, coactivation.
Grober and Buschke test (16 items) (for patients with trasient global amnesia) | Baseline
  Assessement of episodic verbal memory
Brief Visuospatial Memory Test-Revised | Baseline
  Measure of visuospatial memory (for patients with trasient global amnesia)
Forces of the upper limb on the REAplan robot (CIRCUIT, EASY, REACHING) | change between Baseline Day1 and Day3 (acute) + between Baseline Day1 and 3/6 and 12 months post-stroke (subacute - chronic)
  To evaluate the Force of the upper limb after stroke (Newton)
Spectral Arc Lenght on the REAplan robot (CIRCUIT, EASY, REACHING) | change between Baseline Day1 and Day3 (acute) + between Baseline Day1 and 3/6 and 12 months post-stroke (subacute - chronic)
  Movement smoothness quantification
Total distance of the upper limb on the REAplan robot (CIRCUIT, EASY, REACHING) | change between Baseline Day1 and Day3 (acute) + between Baseline Day1 and 3/6 and 12 months post-stroke (subacute - chronic)
  Measure of total distance traveled during the training (cm)
transcranial magnetic stimulation (TMS) | correlation with the measure realized Day 1 with progression of the motor skill learning (change between Baseline Day1 and Day 3)
  Measure of the prediction recovery after stroke

CONTACTS AND LOCATIONS:
Overall Officials: Yves Vandermeeren, MD, PhD, Principal Investigator — UCLouvain IONS
Locations (2):
- Belgium (2):
  - CHU UCL Namur, Yvoir, Namur
  - University Hospital CHU Dinant Godinne UCL, Yvoir

IPD SHARING:
Plan to Share IPD: Yes
the precise IPD plan has to be worked out if an easy and user-friendly solution is available, we intend to make the data available (after anonymisation of personal data).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will become available during thebeggining of the study and for 20 years.
Access Criteria: Login user of the Hospital of CHU UCL Namur -Site Godinne